CLINICAL TRIAL: NCT03911570
Title: Symptomatic Effects of Long-term Crystalline Glucosamine Sulfate Therapy in Hand Osteoarthritis: a Comparative Retrospective Study
Brief Title: Crystalline Glucosamine Sulfate Therapy in Hand Osteoarthritis
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, fioravanti antonella, Symptomatic Effects of Long-term Crystalline Glucosamine Sulfate Therapy in Hand Osteoarthritis: a Comparative Retrospective Study, University of Siena
Other Study IDs: GS-HOA
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Hand Osteoarthritis
MeSH Terms: interventions — Glucosamine; Acetaminophen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Glucosamine Sulfate Group (GS Group): GS Group is treated for at least 6 consecutive months with a single daily dose of 1500 mg of crystalline GS (powder sachets), in addition to conventional therapy.
  Interventions: Drug: Glucosamine Sulfate
- Control Group: Control Group receive only usual care therapy. The conventional therapy includes exercise for HOA and treatment with acetaminophen or oral NSAIDs or COX-2 inhibitors (150 mg Diclofenac tablets, 20 mg Piroxicam tablets, 550 mg Naproxen tablets, 200 mg Aceclofenac, 600 mg Ibuprofen tablets, 200 mg Celecoxib tablets, 60 mg Etoricoxib tablets).
  Interventions: Drug: Glucosamine Sulfate

INTERVENTIONS:
Drug: Glucosamine Sulfate — Therapy with the prescription formulation of crystalline glucosamine sulfate
  Other Names: acetaminophen; non steroidal anti-inflammatory drugs

SUMMARY:
The objective of this study is to retrospectively evaluate the symptomatic effects of crystalline glucosamine sulfate (GS), prescribed for the actually approved indication of knee OA, in addition to conventional therapy, in comparison to the conventional therapy alone in patients with primary hand osteoarthritis (HOA).This is a 6-months retrospective comparative study including patients with concomitant knee and primary HOA, according to the ACR criteria. To be eligible the patients had to present clinical symptoms of hand OA for at least 3 months, defined as global hand pain score superior to 40 mm on a 0-100 Visual Analogue Scale (VAS) and a Functional Index for Hand Osteoarthritis (FIHOA) score of at least 6. Furthermore, the patients have had a radiographic evidence of HOA within the previous 6 months with a Kellgren-Lawrence score of II-III. The participants are stratified into two groups based on whether or not crystalline GS at the daily dose of 1500 mg was added to the conventional therapy for HOA, including exercise, acetaminophen and non steroidal anti-inflammatory drugs (NSAIDs) or cyclo-oxygenase (COX)-2 inhibitors. Primary outcome measures are the difference between the two groups in the change of VAS pain and in the FIHOA, from baseline after 6 months. Secondary outcomes were health assessment questionnaire (HAQ), medical outcomes study 36-item short form (SF-36) and symptomatic drugs consumption.

ELIGIBILITY:
Inclusion Criteria:

* Mono or bilateral primary HOA and concomitant knee OA, according to the American College of Rheumatology (ACR) criteria
* Treatment for at least 6 consecutive months with crystalline GS at the daily dose of 1500 mg in addition to the conventional therapy or with usual care alone.
* HOA symptoms duration for at least 3 months defined as global hand pain score superior to 40 mm on a 0-100 VAS and a FIHOA score of at least 6.
* Radiographic evidence of HOA within the previous 6 months with a radiological score of II-III (using the Kellgren method).

Exclusion Criteria:

* Erosive Osteoarthritis of the hand
* Medical history of any inflammatory joint disease, septic arthritis, previous articular fracture of the concerned joints, monarticular post-traumatic OA of the finger, a history or the presence of any other rheumatic diseases that could cause secondary OA, such as hemochromatosis.
* Ongoing therapy with opioid analgesics and any kind of topical treatment
* Therapy with SYSADOAs other than GS, steroids by any route of administration and intra-articular injection of any joint with hyaluronic acid during the previous 6 months.
* Contraindications or special warnings for GS presented in the data sheet.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants were stratified into two groups based on whether or not (GS Group and Control Group) crystalline GS treatment, prescribed for the actually approved indication of knee OA, was added to the conventional therapy. This stratification was based on regrouping patients with similar clinical characteristics at baseline.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Difference between the two groups in the change of the patient's assessment of global hand pain on a 0- 100 mm Visual Analogue Scale | Basal time; one month; three months; six months
  0-100 mm scale with 0 representing the absence of pain

SECONDARY OUTCOMES:
Difference between the two groups in the change of the Functional Index for Hand Osteoarthritis (FIHOA) score | Basal time; one month; three months; six months
  The FIHOA score represents a quantitative measure of functional disability of the hands; it contains 10 items and is an investigator-administered questionnaire. Patients are asked to answer each item using a four-point Likert scale: 0 = possible without difficulty, 1 = possible with slight difficulty, 2 = possible with considerable difficulty, 3 = impossible; the range of scores is 0-30 and the highest values indicate the worst functionality. The validate Italian version of FIHOA is used for the present study.
Health Assessment Questionnaire (HAQ) | Basal time; one month; three months; six months
  HAQ is a self administered questionnaire developed to measure disability consisting of 8 sections: dressing arising, eating, walking, hygiene, reach, grip, and activities and ranging from 0 to 3 with a higher score corresponding to worse disability
Medical Outcomes Study 36-Item Short Form (SF-36) | Basal time; one month; three months; six months
  SF-36 is a widely used measure of health and wellbeing, including two main domains, mental and physical component summary (MCS and PCS respectively), that investigates 8 different areas of perceived health, such as physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role and mental health. Scores range from "0 to 100" where "0" indicates the worst condition and "100" indicates the best possible condition
NSAIDs and/or acetaminophen consumption | Basal time; one month; three months; six months
  The acetaminophen and NSAIDs/COX-2 inhibitors consumption was calculated asking the patients at each visit the number of tablets taken weekly.

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Unit Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tenti S, Giordano N, Mondanelli N, Giannotti S, Maheu E, Fioravanti A. A retrospective observational study of glucosamine sulfate in addition to conventional therapy in hand osteoarthritis patients compared to conventional treatment alone. Aging Clin Exp Res. 2020 Jun;32(6):1161-1172. doi: 10.1007/s40520-019-01305-4. Epub 2019 Aug 19. PMID 31429006